CLINICAL TRIAL: NCT00475670
Title: An Open-label Study of the Effect of First-line Herceptin Alone or in Combination With a Taxane on Tumor Response and Disease Progression in Patients With Metastatic Breast Cancer Who Relapsed After Receiving Adjuvant Herceptin for HER2-positive Early Breast Cancer
Brief Title: A Study of Herceptin (Trastuzumab) in Women With Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WO17299
Record Dates: First submitted 2007-05-17; First posted 2007-05-21 (Estimated); Results first posted 2014-09-15 (Estimated); Last update posted 2014-09-15 (Estimated); Status verified 2014-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; taxane; Docetaxel; Paclitaxel

ARMS (2):
- Trastuzumab Monotherapy (Active Comparator): Participants received an initial loading dose of 4 milligrams per kilogram (mg/kg) trastuzumab intravenous (i.v.) on Day 1, followed by 2mg/kg i.v. weekly, or an initial loading dose of 8 mg/kg i.v. loading dose on Day 1, followed by 6 mg/kg i.v. every 3 weeks, until disease progression, unacceptable toxicity, withdrawal or death.
  Interventions: Drug: Trastuzumab
- Trastuzumab, Taxane (Experimental): Participant received an initial loading dose of 4 mg/kg trastuzumab i.v. on Day 1, followed by 2mg/kg i.v. weekly, or an initial loading dose of 8 mg/kg i.v. loading dose, followed by 6 mg/kg i.v. every 3 weeks, until disease progression, unacceptable toxicity, withdrawal or death; and concomitant taxane, which is either 100 milligrams per square meter (mg/m2) docetaxel i.v. every 3 weeks, or 75 mg/m2 weekly or 175 mg/m2 every 3 weeks paclitaxel for at least 18 weeks, or more at the discretion of the investigator.
  Interventions: Drug: Trastuzumab; Drug: Taxane (docetaxel or paclitaxel)

INTERVENTIONS:
Drug: Trastuzumab — 4 mg/kg i.v. loading dose on Day 1, followed by 2 mg/kg i.v. weekly; or 8 mg/kg i.v. loading dose, followed by 6 mg/kg i.v. every 3 weeks until disease progression, unacceptable toxicity, withdrawal or death.
  Other Names: Herceptin
Drug: Taxane (docetaxel or paclitaxel) — Docetaxel 100 mg/m2 i.v. every 3 weeks, or paclitaxel administered in a dose of 75 mg/m2 i.v. weekly or 175 mg/m2 i.v. every 3 weeks for at least 18 weeks, or more at the discretion of the investigator. Choice of taxane at the discretion of the investigator. Taxane may be administered at the same time, or 24 hours after, administration of trastuzumab.
  Other Names: Docetaxel; Paclitaxel
  Arms: Trastuzumab, Taxane

SUMMARY:
This 2 arm study will assess the efficacy and safety of intravenous Herceptin with or without a taxane for the first line treatment of metastatic breast cancer in women who have relapsed at least 12 months after a minimum of 10 months of (neo)adjuvant treatment with Herceptin for HER2-positive early breast cancer.Patients will receive either Herceptin monotherapy (loading dose of 4mg/kg iv, followed by weekly doses of 2mg/kg iv, or 8mg/kg loading dose followed by 3-weekly doses of 6mg/kg)or Herceptin + a taxane (docetaxel 100mg/m2 iv every 3 weeks, or paclitaxel 175mg/m2 iv every 3 weeks or 75mg/m2 every week). The anticipated time on study treatment is until disease progression, and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* at least 10 months of Herceptin treatment for HER2-positive early breast cancer;
* metastatic breast cancer >=12 months after discontinuation of Herceptin;
* measurable disease.

Exclusion Criteria:

* previous chemotherapy for metastatic breast cancer;
* brain metastases;
* invasive malignancy other than metastatic breast cancer.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2005-10; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (49):
- Geelong, Victoria, Australia
- Austria (4):
  - Klagenfurt
  - Salzburg
  - Vienna
  - Vöcklabruck
- Belgium (2):
  - Brussels
  - Namur
- Porto Alegre, Rio Grande do Sul, Brazil
- Canada (4):
  - Winnipeg, Manitoba
  - Brampton, Ontario
  - Oshawa, Ontario
  - Greenfield Park, Quebec
- China (4):
  - Beijing
  - Guangzhou
  - Shanghai
  - Wuhan
- Germany (8):
  - Berlin
  - Cologne
  - Düsseldorf
  - Hamburg
  - Krefeld
  - Lemgo
  - München
  - Tübingen
- Hungary (3):
  - Budapest
  - Kecskemét
  - Szeged
- Italy (5):
  - Chieti
  - Genova
  - Roma
  - San Giovanni Rotondo
  - Sassari
- Mérida, Mexico
- Panama City, Panama
- Poland (3):
  - Gdansk
  - Gliwice
  - Lodz
- Russia (3):
  - Kazan'
  - Moscow
  - Saint Petersburg
- Spain (6):
  - Barcelona, Barcelona
  - Jaén, Jaen
  - A Coruña, La Coruña
  - Madrid, Madrid
  - Valencia, Valencia
  - Zaragoza, Zaragoza
- Taiwan (3):
  - Changhua
  - Taipei
  - Taoyuan District

REFERENCES:
- [Derived] Lang I, Bell R, Feng FY, Lopez RI, Jassem J, Semiglazov V, Al-Sakaff N, Heinzmann D, Chang J. Trastuzumab retreatment after relapse on adjuvant trastuzumab therapy for human epidermal growth factor receptor 2-positive breast cancer: final results of the Retreatment after HErceptin Adjuvant trial. Clin Oncol (R Coll Radiol). 2014 Feb;26(2):81-9. doi: 10.1016/j.clon.2013.08.011. Epub 2013 Sep 17. PMID 24051172

RESULTS

PARTICIPANT FLOW:
Groups:
- Trastuzumab Monotherapy: Participants received either an initial loading dose of trastuzumab 4 milligrams per kilogram (mg/kg), intravenously (IV), on Day 1, followed by 2 mg/kg, IV, once per week, or an initial loading dose of 8 mg/kg IV on Day 1, followed by 6 mg/kg IV once every 3 weeks, until disease progression, unacceptable toxicity, withdrawal or death.
- Trastuzumab, Taxane: Participants received either an initial loading dose of trastuzumab 4 mg/kg IV on Day 1, followed by 2 mg/kg IV once per week, or an initial loading dose of 8 mg/kg IV on Day 1, followed by 6 mg/kg IV every 3 weeks, until disease progression, unacceptable toxicity, withdrawal or death. Participants also received one of the following taxanes (at the investigator's discretion) for at least 18 weeks: docetaxel 100 mg/square meter (m^2), IV, once every 3 weeks, OR, paclitaxel 75 mg/m^2, IV, once per week, OR, paclitaxel 175 mg/m^2, IV, once every 3 weeks.
Period: Overall Study
Arm/Group | Trastuzumab Monotherapy | Trastuzumab, Taxane
Started | 3 | 41
Completed | 0 (This cohort was closed prematurely (with only 3 participants) because of enrollment difficulties.) | 0
Not Completed | 3 | 41
Not completed — Death | 0 | 1
Not completed — Lack of Efficacy | 3 | 34
Not completed — Refused treatment | 0 | 2
Not completed — Failure to Return | 0 | 1
Not completed — Other | 0 | 3

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all enrolled participants who received at least one dose of either trastuzumab or taxane.
Groups:
- Trastuzumab Monotherapy: Participants received either an initial loading dose of trastuzumab 4 mg/kg, IV, on Day 1, followed by 2 mg/kg, IV, once per week, or an initial loading dose of 8 mg/kg IV on Day 1, followed by 6 mg/kg IV once every 3 weeks, until disease progression, unacceptable toxicity, withdrawal or death.
- Trastuzumab, Taxane: Participants received either an initial loading dose of trastuzumab 4 mg/kg IV on Day 1, followed by 2 mg/kg IV once per week, or an initial loading dose of 8 mg/kg IV on Day 1, followed by 6 mg/kg IV every 3 weeks, until disease progression, unacceptable toxicity, withdrawal or death. Participants also received one of the following taxanes (at the investigator's discretion) for at least 18 weeks: docetaxel 100 mg/m^2, IV, once every 3 weeks, OR, paclitaxel 75 mg/m^2, IV, once per week, OR, paclitaxel 175 mg/m^2, IV, once every 3 weeks.
- Total: Total of all reporting groups
Arm/Group | Trastuzumab Monotherapy | Trastuzumab, Taxane | Total
Number analyzed (Participants) | 3 | 41 | 44
Age, Continuous [Median (Full Range); unit: years] | 40 [35 to 58] | 54 [31 to 78] | 54 [31 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 41 | 44
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Complete Response (CR) or Partial Response (PR) According to the Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.0 Guidelines
Description: CR was defined for target lesions (TLs) as the disappearance of all lesions, and for nontarget lesions (NTLs) as the disappearance of all nontarget nonmeasurable lesions. PR was defined for TLs as at least a 30 percent (%) decrease from baseline (BL) in the sum of longest diameter (SLD) of TLs. 95% confidence interval for one-sample binomial using Pearson-Clopper method.
Time Frame: Baseline (BL); Day 1 of Weeks 7, 13, 19, 25, 37, and 52, at the last administration of study treatment, every 24 weeks thereafter until disease progression for up to 6 months after the last participant was recruited
Population: FAS; Cohort A (trastuzumab monotherapy) was closed prematurely due to enrollment difficulties. Therefore, Cohort A included only 3 participants and none of the data from these 3 participants were analyzed for any of the specified endpoints.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Trastuzumab Monotherapy | Trastuzumab, Taxane
Number analyzed (Participants) | 0 | 41
percentage of participants |  | 61.0 [48.7 to 80.4]

2. Secondary Outcome: Duration of Response - Percentage of Participants With Progressive Disease or Death
Description: Duration of response was defined as the time from first confirmed CR or PR until death or progressive disease (PD). For TLs, PD was defined as at least a 20% increase in the SLD of the TL, taking as reference the smallest SLD recorded since the beginning of treatment or the appearance of one or more new lesions. For NTLs, PD was defined as the appearance of one or more new lesions or unequivocal progression of existing non target non-measurable lesions. Participants were censored at the date of the last tumor assessment.
Time Frame: BL, Day 1 of Weeks 7, 13, 19, 25, 37, and 52, at the last administration of study treatment, every 24 weeks thereafter until disease progression for up to 6 months after the last participant was recruited
Population: FAS. Duration of response was assessed in participants with a best overall response of CR or PR. Cohort A (trastuzumab monotherapy) was closed prematurely due to enrollment difficulties. Therefore, Cohort A included only 3 participants and none of the data from these 3 participants were analyzed for any of the specified endpoints.
Measure: Number; unit: percentage of participants
Arm/Group | Trastuzumab Monotherapy | Trastuzumab, Taxane
Number analyzed (Participants) | 0 | 25
percentage of participants |  | 88.0

3. Secondary Outcome: Duration of Response
Description: The time, in months, from when the response (CR or PR) was first noted until the date of documented PD, death, or withdrawal, whichever occurred first. Participants were censored at the date of the last tumor assessment.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab Monotherapy | Trastuzumab, Taxane
Number analyzed (Participants) | 0 | 25
months |  | 8.0 [5 to 15]

4. Secondary Outcome: Progression-free Survival (PFS) - Percentage of Participants With Progressive Disease
Description: PFS was defined as the time from day of first study drug infusion until death or PD. Participants were censored at the date of the last tumor assessment.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Trastuzumab Monotherapy | Trastuzumab, Taxane
Number analyzed (Participants) | 0 | 41
percentage of participants |  | 87.8

5. Secondary Outcome: Progression-Free Survival
Description: The time, in months, from BL to PFS event.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab Monotherapy | Trastuzumab, Taxane
Number analyzed (Participants) | 0 | 41
months |  | 8.0 [6 to 11]

6. Secondary Outcome: Percentage of Participants With Treatment Failure
Description: Treatment failure was defined as the time from first study drug infusion to failure. Failure was defined as any of the following: PD, death, withdrawal due to adverse event (AE) or lab abnormality, or refusal of treatment. Participants were censored at the last date recorded in the case report form (CRF) or the date of withdrawal.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Trastuzumab Monotherapy | Trastuzumab, Taxane
Number analyzed (Participants) | 0 | 41
percentage of participants |  | 95.1

7. Secondary Outcome: Time to Treatment Failure
Description: The time, in months, from BL to treatment failure.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab Monotherapy | Trastuzumab, Taxane
Number analyzed (Participants) | 0 | 41
months |  | 8.0 [6 to 11]

8. Secondary Outcome: Percentage of Participants With Clinical Benefit According to RECIST Guidelines
Description: Clinical benefit was defined as stable disease (SD) for 6 months or longer, or a confirmed overall response of CR or PR. For TLs, SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest SLD since the beginning of treatment. For NTLs, SD was synonymous with incomplete response and defined as the persistence of one or more NTLs and/or maintenance of tumor marker level above the normal limits.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Trastuzumab Monotherapy | Trastuzumab, Taxane
Number analyzed (Participants) | 0 | 41
percentage of participants |  | 70.7 [54.5 to 83.9]

9. Secondary Outcome: Overall Survival - Percentage of Participants Who Died
Description: OS was defined as the time from the date of enrollment to the date of death due to any cause. Participants were censored at the last date recorded in the CRF.
Time Frame: BL, Day 1 of Weeks 1, 4, 7, 10, 13, 16, 19, 25, 37, and 5 at the last administration of study treatment, every 24 weeks thereafter until disease progression or death, yearly thereafter up to 2 years after cessation of recruitment
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Trastuzumab Monotherapy | Trastuzumab, Taxane
Number analyzed (Participants) | 0 | 41
percentage of participants |  | 63.4

10. Secondary Outcome: Overall Survival
Description: The time, in months, from BL to death due to any cause.
Time Frame: BL, Day 1 of Weeks 1, 4, 7, 10, 13, 16, 19, 25, 37, and 52 at the last administration of study treatment, every 24 weeks thereafter until disease progression or death, yearly thereafter up to 2 years after cessation of recruitment
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab Monotherapy | Trastuzumab, Taxane
Number analyzed (Participants) | 0 | 41
months |  | 25.0 [16 to 33]

ADVERSE EVENTS:
Time Frame: Adverse events and serious adverse events were recorded from study start to 28 days after the last dose of study drug. Serious adverse events that were related to study medication or were cardiac are reported until 2 years after enrollment.
Description: The safety analysis population included all participants who received at least 1 dose of either trastuzumab or taxane.
Arm/Group | Trastuzumab Monotherapy | Trastuzumab, Taxane
Serious Adverse Events (participants affected / at risk) | 0/3 | 6/41
Other Adverse Events (participants affected / at risk) | 3/3 | 36/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab Monotherapy (N=3) | Trastuzumab, Taxane (N=41)
Bacterial Infection (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Sudden Death (General disorders) | 0 | 1
Lymphoedema (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab Monotherapy (N=3) | Trastuzumab, Taxane (N=41)
Neutropenia (Blood and lymphatic system disorders) | 0 | 5
Lacrimation increased (Eye disorders) | 0 | 4
Abdominal pain (Gastrointestinal disorders) | 0 | 4
Diarrhoea (Gastrointestinal disorders) | 0 | 13
Dyspepsia (Gastrointestinal disorders) | 0 | 3
Nausea (Gastrointestinal disorders) | 0 | 6
Stomatitis (Gastrointestinal disorders) | 0 | 4
Vomiting (Gastrointestinal disorders) | 0 | 5
Asthenia (General disorders) | 0 | 6
Fatigue (General disorders) | 0 | 10
Oedema peripheral (General disorders) | 1 | 7
Pyrexia (General disorders) | 1 | 6
Bronchitis (Infections and infestations) | 0 | 4
Nasopharyngitis (Infections and infestations) | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 6
Headache (Nervous system disorders) | 1 | 3
Neuropathy peripheral (Nervous system disorders) | 0 | 3
Paraesthesia (Nervous system disorders) | 0 | 4
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 13
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 3
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 7
Rash (Skin and subcutaneous tissue disorders) | 0 | 6
Urinary tract infection (Infections and infestations) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Cohort A (trastuzumab monotherapy) was closed prematurely due to enrollment difficulties. Therefore, Cohort A included only 3 participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.